CLINICAL TRIAL: NCT03538938
Title: Improving Quitline Support Study: Optimizing Remotely Delivered Smoking Cessation Services for Low-Income Smokers
Brief Title: Improving Quitline Support Study
Acronym: IQS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: George Washington University (Other); Consumer Wellness Solutions (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-0553; Protocol Version 11/18/2020 (Other: UW Madison); 1R01CA218156-01 (NIH); A534252 (Other: UW Madison); SMPH\MEDICINE\TOBACCO RE (Other: UW Madison); UW20069 (Other: UW Madison)
Record Dates: First submitted 2018-05-03; First posted 2018-05-29 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Tobacco Use Cessation
Keywords: Smoking; Smoking cessation; Quitline; Nicotine Replacement Therapy; SmokefreeTXT text messages; Financial incentives
MeSH Terms: conditions — Tobacco Use Cessation; Smoking; Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Four-factor fully-crossed factorial design
Who Masked: Outcomes Assessor
Masking Description: Research staff who conduct follow-up interviews and verification will be blind to study condition and will not have access to other participant data (e.g., smoking history) prior to the end of data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (16):
- 1-Call, Patch, SmokefreeTXT, Financial Incentive (Experimental): Participants will receive the following treatment combination: 1-Call Quitline Counseling, two weeks of Nicotine Patch, instruction in enrolling in SmokefreeTXT, and Financial Incentives for Treatment Engagement. The proactive counseling call will last approximately 20 minutes. The Nicotine Patch treatment will consist of a two week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD). SmokefreeTXT text messaging in support of cessation will consist of 6-8 weeks of text messages (up to 5 messages per day for up to two weeks prior to the target quit day and for six weeks following the target quit day). Financial Incentives for treatment engagement are for completing the counseling call and for staying enrolled in the SmokefreeTXT program for six weeks.
  Interventions: Behavioral: 1-Call Quitline Counseling; Drug: Nicotine patch; Behavioral: SmokefreeTXT; Behavioral: Financial Incentives for Treatment Engagement
- 1-Call, Patch, SmokefreeTXT, No Financial Incentive (Experimental): Participants will receive the following treatment combination: 1-Call Quitline Counseling, two weeks of Nicotine Patch, instruction in enrolling in SmokefreeTXT, No Financial Incentives for Treatment Engagement. The proactive counseling call will last approximately 20 minutes. The Nicotine Patch treatment will consist of a two week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD). SmokefreeTXT text messaging in support of cessation will consist of 6-8 weeks of text messages (up to 5 messages per day for up to two weeks prior to the target quit day and for six weeks following the target quit day). Financial Incentives for treatment engagement will not be offered.
  Interventions: Behavioral: 1-Call Quitline Counseling; Drug: Nicotine patch; Behavioral: SmokefreeTXT; Behavioral: No Financial Incentives for Treatment Engagement
- 1-Call, Patch, No SmokefreeTXT, Financial Incentive (Experimental): Participants will receive the following treatment combination: 1-Call Quitline Counseling, two weeks of Nicotine Patch, No SmokefreeTXT, and Financial Incentives for Treatment Engagement. The proactive counseling call will last approximately 20 minutes. The Nicotine Patch treatment will consist of a two week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD). SmokefreeTXT text messaging in support of cessation will not be offered proactively. Financial Incentives for treatment engagement are for completing the counseling call.
  Interventions: Behavioral: 1-Call Quitline Counseling; Drug: Nicotine patch; Behavioral: No SmokefreeTXT; Behavioral: Financial Incentives for Treatment Engagement
- 1-Call, Patch, No SmokefreeTXT, No Financial Incentive (Experimental): Participants will receive the following treatment combination: 1-Call Quitline Counseling, two weeks of Nicotine Patch, No SmokeFreeTXT, and No Financial Incentives for Treatment Engagement. The proactive counseling call will last approximately 20 minutes. The Nicotine Patch treatment will consist of a two week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD). SmokefreeTXT text messaging in support of cessation will not be offered proactively. Financial Incentives for treatment engagement will not be offered.
  Interventions: Behavioral: 1-Call Quitline Counseling; Drug: Nicotine patch; Behavioral: No SmokefreeTXT; Behavioral: No Financial Incentives for Treatment Engagement
- 1-Call, Patch+Loz, SmokefreeTXT, Financial Incentive (Experimental): Participants will receive the following: 1-Call Quitline Counseling, 4 weeks of Nicotine Patch and Nicotine Lozenges, instruction in enrolling in SmokefreeTXT, and Financial Incentives for Treatment Engagement. The proactive counseling call will last approximately 20 minutes. Patch treatment will consist of a 4 week supply of over-the-counter nicotine patches (21 mg if smoking 10 or more cigarettes per day (CPD); 14 mg if smoking fewer than 10 CPD); Lozenge treatment will consist of a four week supply of over-the-counter nicotine lozenges (2-mg dose for those who do not smoke within 30 minutes of waking; 4-mg dose for those who smoke within 30 minutes of waking). SmokefreeTXT will consist of 6-8 weeks of text messages (up to 5 messages per day for up to two weeks prior to the target quit day [TQD] and for 6 weeks following the TQD). The Financial Incentives are for completing the counseling call and for staying enrolled in the SmokefreeTXT program for 6 weeks.
  Interventions: Behavioral: 1-Call Quitline Counseling; Drug: Nicotine Patch and Nicotine Lozenge; Behavioral: SmokefreeTXT; Behavioral: Financial Incentives for Treatment Engagement
- 1-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive (Experimental): Participants will receive the following treatment combination: 1-Call Quitline Counseling, four weeks of Nicotine Patch and Nicotine Lozenges, instruction in enrolling in SmokefreeTXT, and No Financial Incentives for Treatment Engagement. The proactive counseling call will last approximately 20 minutes. Nicotine Patch treatment will consist of a 4-week supply of over-the-counter nicotine patches (21 mg if smoking 10 or more cigarettes per day (CPD); 14 mg if smoking fewer than 10 CPD); Lozenge treatment will consist of a 4-week supply of over-the-counter nicotine lozenges (2-mg dose for those who do not smoke within 30 minutes of waking; 4-mg dose for those who smoke within 30 minutes of waking). SmokefreeTXT text messaging in support of cessation will consist of 6-8 weeks of text messages (up to 5 messages per day for up to 2 weeks prior to the target quit day and for six weeks following the target quit day). Financial Incentives for treatment engagement will not be offered.
  Interventions: Behavioral: 1-Call Quitline Counseling; Drug: Nicotine Patch and Nicotine Lozenge; Behavioral: SmokefreeTXT; Behavioral: No Financial Incentives for Treatment Engagement
- 1-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive (Experimental): Participants will receive the following treatment combination: 1-Call Quitline Counseling, four weeks of Nicotine Patch and Nicotine Lozenges, No SmokefreeTXT, and Financial Incentives for Treatment Engagement. The proactive counseling call will last approximately 20 minutes. The Nicotine Patch treatment will consist of a four week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD); Lozenge treatment will consist of a four week supply of over-the-counter nicotine lozenges (2-mg dose for those who do not smoke within 30 minutes of waking; 4-mg dose for those who smoke within 30 minutes of waking). No SmokefreeTXT text messaging in support of cessation will be offered proactively. The Financial Incentives for treatment engagement are for completing the counseling call.
  Interventions: Behavioral: 1-Call Quitline Counseling; Drug: Nicotine Patch and Nicotine Lozenge; Behavioral: No SmokefreeTXT; Behavioral: Financial Incentives for Treatment Engagement
- 1-Call, Patch+Loz, No SmokefreeTXT, No Financial Incentive (Experimental): Participants will receive the following treatment combination: 1-Call Quitline Counseling, four weeks of Nicotine Patch and Nicotine Lozenges, No SmokefreeTXT, and No Financial Incentives for Treatment Engagement. The proactive counseling call will last approximately 20 minutes. The Patch treatment will consist of a four week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD); Lozenge treatment will consist of a four week supply of over-the-counter nicotine lozenges (2-mg dose for those who do not smoke within 30 minutes of waking; 4-mg dose for those who smoke within 30 minutes of waking). SmokefreeTXT text messaging in support of cessation will not be offered proactively. Financial Incentives for treatment engagement will not be offered.
  Interventions: Behavioral: 1-Call Quitline Counseling; Drug: Nicotine Patch and Nicotine Lozenge; Behavioral: No SmokefreeTXT; Behavioral: No Financial Incentives for Treatment Engagement
- 4-Call, Patch, SmokefreeTXT, Financial Incentive (Experimental): Participants will receive the following treatment combination:4-Call Quitline Counseling, two weeks of Nicotine Patch, instruction in enrolling in SmokefreeTXT, and Financial Incentives for Treatment Engagement. Each of the proactive counseling calls will last approximately 20 minutes. The Nicotine Patch treatment will consist of a two week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD). SmokefreeTXT text messaging in support of cessation will consist of 6-8 weeks of text messages (up to 5 messages per day for up to two weeks prior to the target quit day and for six weeks following the target quit day). The Financial Incentives for treatment engagement are for completing each of the four counseling calls and for staying enrolled in the SmokefreeTXT program for six weeks.
  Interventions: Behavioral: 4-Call Quitline Counseling; Drug: Nicotine patch; Behavioral: SmokefreeTXT; Behavioral: Financial Incentives for Treatment Engagement
- 4-Call, Patch, SmokefreeTXT, No Financial Incentive (Experimental): Participants will receive the following treatment combination: 4-Call Quitline Counseling, two weeks of Nicotine Patch, instruction in enrolling in SmokefreeTXT, and No Financial Incentives for Treatment Engagement. Each of the proactive counseling calls will last approximately 20 minutes. The Nicotine Patch treatment will consist of a two week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD). SmokefreeTXT text messaging in support of cessation will consist of 6-8 weeks of text messages (up to 5 messages per day for up to two weeks prior to the target quit day and for six weeks following the target quit day). Financial Incentives for treatment engagement will not be offered.
  Interventions: Behavioral: 4-Call Quitline Counseling; Drug: Nicotine patch; Behavioral: SmokefreeTXT; Behavioral: No Financial Incentives for Treatment Engagement
- 4-Call, Patch, No SmokefreeTXT, Financial Incentive (Experimental): Participants will receive the following treatment combination: 4-Call Quitline Counseling, two weeks of Nicotine Patch, No SmokefreeTXT, and Financial Incentives for Treatment Engagement. Each of the proactive counseling calls will last approximately 20 minutes. The Nicotine Patch treatment will consist of a two week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD). SmokefreeTXT text messaging in support of cessation will not be offered proactively. The Financial Incentives for treatment engagement are for completing each of the four counseling calls.
  Interventions: Behavioral: 4-Call Quitline Counseling; Drug: Nicotine patch; Behavioral: No SmokefreeTXT; Behavioral: Financial Incentives for Treatment Engagement
- 4-Call, Patch, No SmokefreeTXT, No Financial Incentive (Experimental): Participants will receive the following treatment combination: 4-Call Quitline Counseling, two weeks of Nicotine Patch, No SmokefreeTXT, and No Financial Incentives for Treatment Engagement. Each of the proactive counseling calls will last approximately 20 minutes. The Nicotine Patch treatment will consist of a two week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD). SmokefreeTXT text messaging in support of cessation will not be offered proactively. Financial Incentives for treatment engagement will not be offered.
  Interventions: Behavioral: 4-Call Quitline Counseling; Drug: Nicotine patch; Behavioral: No SmokefreeTXT; Behavioral: No Financial Incentives for Treatment Engagement
- 4-Call, Patch+Loz, SmokefreeTXT, Financial Incentive (Experimental): Participants will receive: 4-Call Quitline Counseling, 4 weeks of Nicotine Patch and Nicotine Lozenges, instruction in enrolling in SmokefreeTXT, and Financial Incentives for Treatment Engagement. Each counseling call will last approximately 20 min. Patch treatment will consist of a 4 week supply of over-the-counter (OTC) nicotine patches (21 mg for if smoking 10 or more cigarettes per day (CPD); 14 mg if smoking fewer than 10 CPD); Lozenge treatment will consist of a 4 week supply of OTC nicotine lozenges (2-mg dose for those who do not smoke within 30 min of waking; 4-mg dose for those who smoke within 30 min of waking). SmokefreeTXT in support of cessation will consist of 6-8 weeks of text messages (up to 5 messages per day for up to 2 weeks prior to the target quit day [TQD] and for 6 weeks following the TQD). Financial Incentives are for completing each of the 4 counseling calls and for staying enrolled in SmokefreeTXT for 6 weeks.
  Interventions: Behavioral: 4-Call Quitline Counseling; Drug: Nicotine Patch and Nicotine Lozenge; Behavioral: SmokefreeTXT; Behavioral: Financial Incentives for Treatment Engagement
- 4-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive (Experimental): Participants will receive the following treatment combination: 4-Call Quitline Counseling, four weeks of Nicotine Patch and Nicotine Lozenges, instruction in enrolling in SmokefreeTXT, and No Financial Incentives for Treatment Engagement. Each of the proactive counseling calls will last approximately 20 minutes. The Patch treatment will consist of a 4-week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD); Lozenge treatment will consist of a 4-week supply of over-the-counter nicotine lozenges (2-mg dose for those who do not smoke within 30 minutes of waking; 4-mg dose for those who smoke within 30 minutes of waking). SmokefreeTXT in support of cessation will consist of 6-8 weeks of text messages (up to 5 messages per day for up to 2 weeks prior to the target quit day and for 6 weeks following the target quit day). Financial Incentives for treatment engagement will not be offered.
  Interventions: Behavioral: 4-Call Quitline Counseling; Drug: Nicotine Patch and Nicotine Lozenge; Behavioral: SmokefreeTXT; Behavioral: No Financial Incentives for Treatment Engagement
- 4-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive (Experimental): Participants will receive the following treatment combination: 4-Call Quitline Counseling, four weeks of Nicotine Patch and Nicotine Lozenge, No SmokefreeTXT, and Financial Incentives for Treatment Engagement. Each of the proactive counseling calls will last approximately 20 minutes. The Nicotine Patch treatment will consist of a four week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD); Lozenge treatment will consist of a four week supply of over-the-counter nicotine lozenges (2-mg dose for those who do not smoke within 30 minutes of waking; 4-mg dose for those who smoke within 30 minutes of waking). SmokefreeTXT text messaging in support of cessation will not be offered proactively. The Financial Incentives for treatment engagement are for completing each of the four counseling calls.
  Interventions: Behavioral: 4-Call Quitline Counseling; Drug: Nicotine Patch and Nicotine Lozenge; Behavioral: No SmokefreeTXT; Behavioral: Financial Incentives for Treatment Engagement
- 4-Call, Patch+Loz, No SmokefreeTXT,No Financial Incentive (Experimental): Participants will receive the following treatment combination: 4-Call Quitline Counseling, four weeks of Nicotine Patch and Nicotine Lozenges, No SmokefreeTXT, and No Financial Incentives for Treatment Engagement. Each of the proactive counseling calls will last approximately 20 minutes. The Patch treatment will consist of a four week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD); Lozenge treatment will consist of a four week supply of over-the-counter nicotine lozenges (2-mg dose for those who do not smoke within 30 minutes of waking; 4-mg dose for those who smoke within 30 minutes of waking). SmokefreeTXT in support of cessation will not be offered proactively. Financial Incentives for treatment engagement will not be offered.
  Interventions: Behavioral: 4-Call Quitline Counseling; Drug: Nicotine Patch and Nicotine Lozenge; Behavioral: No SmokefreeTXT; Behavioral: No Financial Incentives for Treatment Engagement

INTERVENTIONS:
Behavioral: 1-Call Quitline Counseling — The 1-Call Quitline Counseling will be provided by the Wisconsin Tobacco Quit Line (WTQL) and consists of 1 proactive call using a standard, evidence-based protocol lasting approximately 20 minutes; ad hoc calls that are initiated by the participant are also available.
  Arms: 1-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive; 1-Call, Patch+Loz, No SmokefreeTXT, No Financial Incentive; 1-Call, Patch+Loz, SmokefreeTXT, Financial Incentive; 1-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive; 1-Call, Patch, No SmokefreeTXT, Financial Incentive; 1-Call, Patch, No SmokefreeTXT, No Financial Incentive; 1-Call, Patch, SmokefreeTXT, Financial Incentive; 1-Call, Patch, SmokefreeTXT, No Financial Incentive
Behavioral: 4-Call Quitline Counseling — The 4-Call Quitline Counseling will be provided by the Wisconsin Tobacco Quit Line (WTQL) and consists of 4 proactive calls that use a standard, evidence-based protocol with each call lasting approximately 20 minutes; ad hoc calls that are initiated by the participant are also available.
  Arms: 4-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive; 4-Call, Patch+Loz, No SmokefreeTXT,No Financial Incentive; 4-Call, Patch+Loz, SmokefreeTXT, Financial Incentive; 4-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive; 4-Call, Patch, No SmokefreeTXT, Financial Incentive; 4-Call, Patch, No SmokefreeTXT, No Financial Incentive; 4-Call, Patch, SmokefreeTXT, Financial Incentive; 4-Call, Patch, SmokefreeTXT, No Financial Incentive
Drug: Nicotine patch — Nicotine Patch treatment will consist of a two week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD).
  Arms: 1-Call, Patch, No SmokefreeTXT, Financial Incentive; 1-Call, Patch, No SmokefreeTXT, No Financial Incentive; 1-Call, Patch, SmokefreeTXT, Financial Incentive; 1-Call, Patch, SmokefreeTXT, No Financial Incentive; 4-Call, Patch, No SmokefreeTXT, Financial Incentive; 4-Call, Patch, No SmokefreeTXT, No Financial Incentive; 4-Call, Patch, SmokefreeTXT, Financial Incentive; 4-Call, Patch, SmokefreeTXT, No Financial Incentive
Drug: Nicotine Patch and Nicotine Lozenge — The Nicotine Patch treatment will consist of a four week supply of over-the-counter nicotine patches (21 mg for those who smoke 10 or more cigarettes per day (CPD); 14 mg for those who smoke fewer than 10 CPD); the Nicotine Lozenge treatment will consist of a four week supply of over-the-counter nicotine lozenges (2-mg dose for those who do not smoke within 30 minutes of waking; 4-mg dose for those who smoke within 30 minutes of waking).
  Arms: 1-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive; 1-Call, Patch+Loz, No SmokefreeTXT, No Financial Incentive; 1-Call, Patch+Loz, SmokefreeTXT, Financial Incentive; 1-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive; 4-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive; 4-Call, Patch+Loz, No SmokefreeTXT,No Financial Incentive; 4-Call, Patch+Loz, SmokefreeTXT, Financial Incentive; 4-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive
Behavioral: SmokefreeTXT — SmokefreeTXT support is a national program offered at no cost to users (apart from data/minute costs charged by cellular providers about which enrollees are advised at enrollment) and is sponsored by the National Cancer Institute. This program sends up to 5 messages per day for up to 2 weeks prior to the target quit day and 6 weeks following the target quit day (total duration may be longer if participants elect to change the target quit day). The text messages offer tips to help enrollees achieve their goal of quitting smoking and offer real-time interactive tips when participants text in responses indicating cravings, negative moods, or slips. Participants have the option to reset quit dates and have the option to unsubscribe at any time by texting STOP to the program.
  Arms: 1-Call, Patch+Loz, SmokefreeTXT, Financial Incentive; 1-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive; 1-Call, Patch, SmokefreeTXT, Financial Incentive; 1-Call, Patch, SmokefreeTXT, No Financial Incentive; 4-Call, Patch+Loz, SmokefreeTXT, Financial Incentive; 4-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive; 4-Call, Patch, SmokefreeTXT, Financial Incentive; 4-Call, Patch, SmokefreeTXT, No Financial Incentive
Behavioral: No SmokefreeTXT — Proactive information about enrolling in adjunctive SmokefreeTXT text messaging support is not offered.
  Arms: 1-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive; 1-Call, Patch+Loz, No SmokefreeTXT, No Financial Incentive; 1-Call, Patch, No SmokefreeTXT, Financial Incentive; 1-Call, Patch, No SmokefreeTXT, No Financial Incentive; 4-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive; 4-Call, Patch+Loz, No SmokefreeTXT,No Financial Incentive; 4-Call, Patch, No SmokefreeTXT, Financial Incentive; 4-Call, Patch, No SmokefreeTXT, No Financial Incentive
Behavioral: Financial Incentives for Treatment Engagement — Incentives for treatment engagement are for each counseling session and for staying enrolled in SmokefreeTXT for six weeks. These incentives are designed to bolster motivation to stay engaged in treatment and to offset the costs and effort of treatment engagement (in terms of cell phone minutes).
  Arms: 1-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive; 1-Call, Patch+Loz, SmokefreeTXT, Financial Incentive; 1-Call, Patch, No SmokefreeTXT, Financial Incentive; 1-Call, Patch, SmokefreeTXT, Financial Incentive; 4-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive; 4-Call, Patch+Loz, SmokefreeTXT, Financial Incentive; 4-Call, Patch, No SmokefreeTXT, Financial Incentive; 4-Call, Patch, SmokefreeTXT, Financial Incentive
Behavioral: No Financial Incentives for Treatment Engagement — No Financial Incentives for Treatment Engagement are offered.
  Arms: 1-Call, Patch+Loz, No SmokefreeTXT, No Financial Incentive; 1-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive; 1-Call, Patch, No SmokefreeTXT, No Financial Incentive; 1-Call, Patch, SmokefreeTXT, No Financial Incentive; 4-Call, Patch+Loz, No SmokefreeTXT,No Financial Incentive; 4-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive; 4-Call, Patch, No SmokefreeTXT, No Financial Incentive; 4-Call, Patch, SmokefreeTXT, No Financial Incentive

SUMMARY:
This study seeks to evaluate ways to improve outcomes for low-education, uninsured or Medicaid-eligible smokers who do not successfully quit with standard telephone quit line treatment. The study will use an efficient factorial study design to evaluate four evidence-based strategies to improve follow-up care offered by the Wisconsin Tobacco Quit Line (WTQL) to socioeconomically disadvantaged callers who report smoking four months following initial WTQL treatment comprising a single counseling call and 2-week supply of a single nicotine replacement therapy. These strategies include: increasing the intensity of nicotine replacement medication (among those medically cleared to use such medications), increasing the intensity of WTQL counseling, helping callers enroll in an evidence-based smoking cessation texting support program (SmokefreeTXT), and offering moderate financial incentives for engagement in counseling and SmokefreeTXT.

DETAILED DESCRIPTION:
This study seeks to evaluate ways to improve outcomes for low-education, uninsured or Medicaid-eligible smokers who do not successfully quit with standard telephone quit line treatment. The study will use an efficient factorial study design to evaluate four evidence-based strategies to improve follow-up care offered by the Wisconsin Tobacco Quit Line (WTQL) to socioeconomically disadvantaged callers who report smoking four months following initial WTQL treatment comprising a single counseling call and 2-week supply of a single nicotine replacement therapy. The four factors (strategies) to be studied include: (1) Quit line counseling intensity (1 vs 4 proactive calls); (2) Nicotine replacement therapy (NRT) intensity (Patch for 2 weeks vs Patch+Lozenge for 4 weeks); (3) SmokefreeTXT text messages (proactive enrollment vs none); and (4) financial incentives for treatment engagement (vs none). The study design is a fully-crossed 4-factor factorial design. The primary aim is: Assessment of the main and interactive effects of the four treatment factors on biochemically-confirmed 7-day point-prevalence abstinence at the 6-month followup. Secondary aims include testing: (1) self-reported abstinence at 12 weeks post-quit; (2) continuous abstinence between 1 and 6 months; (3) cost-effectiveness; and (4) moderators of treatment engagement and mediators of treatment effectiveness on 6-month abstinence.

ELIGIBILITY:
Inclusion Criteria:

1. Uninsured, covered by BadgerCareWisconsin or another Medicaid program, or has no more than a high school education
2. Lives in Wisconsin
3. Age 18 or older
4. English speaking
5. Must provide a unique telephone number not already registered in the Wisconsin Tobacco Quit Line (WTQL) database for this study (to prevent duplicate enrollment and to ensure that only one person per household enrolls)
6. Must have completed standard WTQL treatment including at least one counseling call 2.5-18 months prior to study recruitment
7. Reported smoking at least 6 of the last 7 days at the WTQL follow-up enrollment call (2.5-18 months after completing standard WTQL treatment), with at least 5 cigarettes smoked on 1 or more days
8. Willing to set a new quit day within 2 weeks

Exclusion Criteria:

1. Pregnancy, breastfeeding, or planning to become pregnant in the next 6 months at the time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1316 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E. McCarthy, PhD, Principal Investigator — University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health
Locations (1):
- Wisconsin Tobacco Quit Line (service provided by Free & Clear, Inc.), Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The University of Wisconsin Center for Tobacco Research and Intervention (UW-CTRI) is committed to making final research datasets available to the scientific community in a timely fashion in accord with general NIH policy. The following are the main types of data that will be generated by this grant:
  * Behavioral, health, and economic data and outcomes for all participants in the primary research.
  * Data on individual differences and risk factors for treatment acceptance, smoking cessation outcomes, and response to cessation treatments.
  In accord with Institutional Review Board (IRB) policies, the UW-CTRI will act under its own auspices as the hub for making de-identified data available. The PI will make the set of final de-identified datasets available by request from other researchers in a timely manner.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified data will be available 1 year after final data collection.
Access Criteria: Researchers who desire access to study data must submit a Data Use Proposal to the PI.
URL: http://www.ctri.wisc.edu

REFERENCES:
- [Derived] Kaye JT, Kirsch JA, Bolt DM, Kobinsky KH, Vickerman KA, Mullis K, Fraser DL, Baker TB, Fiore MC, McCarthy DE. Tobacco Quitline Retreatment Interventions Among Adults With Socioeconomic Disadvantage: A Factorial Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2443044. doi: 10.1001/jamanetworkopen.2024.43044. PMID 39504025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1316 of the target 1408 participants were recruited between June 2018 and January 2023
Groups:
- 1-Call, Patch, SmokefreeTXT, Financial Incentive: Participants received: 1 quitline counseling call, 2 weeks of nicotine patch, SmokefreeTXT information, and financial incentives for treatment engagement
- 1-Call, Patch, SmokefreeTXT, No Financial Incentive: Participants received: 1 quitline counseling call, 2 weeks of nicotine patch, SmokefreeTXT information, and no financial incentives for treatment engagement
- 1-Call, Patch, No SmokefreeTXT, Financial Incentive: Participants received: 1 quitline counseling call, 2 weeks of nicotine patch, no SmokefreeTXT information, and financial incentives for treatment
- 1-Call, Patch, No SmokefreeTXT, No Financial Incentive: Participants received: 1 quitline counseling call, 2 weeks of nicotine patch, no SmokefreeTXT information, and no financial incentives for treatment engagement
- 1-Call, Patch+Loz, SmokefreeTXT, Financial Incentive: Participants received: 1 quitline counseling call, 4 weeks of nicotine patch and nicotine lozenges, SmokefreeTXT information, and financial incentives for treatment engagement
- 1-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive: Participants received: 1 quitline counseling call, 4 weeks of nicotine patch and nicotine lozenges, SmokefreeTXT information, and no financial incentives for treatment engagement
- 1-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive: Participants received: 1 quitline counseling call, 4 weeks of nicotine patch and nicotine lozenges, no SmokefreeTXT information, and financial incentives for treatment engagement
- 1-Call, Patch+Loz, No SmokefreeTXT, No Financial Incentive: Participants received: 1 quitline counseling call, 4 weeks of nicotine patch and nicotine lozenges, no SmokefreeTXT information, and no financial incentives for treatment engagement
- 4-Call, Patch, SmokefreeTXT, Financial Incentive: Participants received: 4 quitline counseling calls, 2 weeks of nicotine patch, SmokefreeTXT information, and financial incentives for treatment engagement
- 4-Call, Patch, SmokefreeTXT, No Financial Incentive: Participants received: 4 quitline counseling calls, 2 weeks of nicotine patch, SmokefreeTXT information, and no financial incentives for treatment engagement
- 4-Call, Patch, No SmokefreeTXT, Financial Incentive: Participants received: 4 quitline counseling calls, 2 weeks of nicotine patch, no SmokefreeTXT information, and financial incentives for treatment engagement
- 4-Call, Patch, No SmokefreeTXT, No Financial Incentive: Participants received: 4 quitline counseling calls, 2 weeks of nicotine patch, no SmokefreeTXT information, and no financial incentives for treatment engagement
- 4-Call, Patch+Loz, SmokefreeTXT, Financial Incentive: Participants received: 4 quitline counseling calls, 4 weeks of nicotine patch and nicotine lozenge, SmokefreeTXT information, and financial incentives for treatment engagement
- 4-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive: Participants received: 4 quitline counseling calls, 4 weeks of nicotine patch and nicotine lozenge, SmokefreeTXT information, and no financial incentives for treatment engagement
- 4-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive: Participants received: 4 quitline counseling calls, 4 weeks of nicotine patch and nicotine lozenge, no SmokefreeTXT information, and financial incentives for treatment engagement
- 4-Call, Patch+Loz, No SmokefreeTXT,No Financial Incentive: Participants received: 4 quitline counseling calls, 4 weeks of nicotine patch and nicotine lozenge, no SmokefreeTXT information, and no financial incentives for treatment engagement
Period: Overall Study
Arm/Group | 1-Call, Patch, SmokefreeTXT, Financial Incentive | 1-Call, Patch, SmokefreeTXT, No Financial Incentive | 1-Call, Patch, No SmokefreeTXT, Financial Incentive | 1-Call, Patch, No SmokefreeTXT, No Financial Incentive | 1-Call, Patch+Loz, SmokefreeTXT, Financial Incentive | 1-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive | 1-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive | 1-Call, Patch+Loz, No SmokefreeTXT, No Financial Incentive | 4-Call, Patch, SmokefreeTXT, Financial Incentive | 4-Call, Patch, SmokefreeTXT, No Financial Incentive | 4-Call, Patch, No SmokefreeTXT, Financial Incentive | 4-Call, Patch, No SmokefreeTXT, No Financial Incentive | 4-Call, Patch+Loz, SmokefreeTXT, Financial Incentive | 4-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive | 4-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive | 4-Call, Patch+Loz, No SmokefreeTXT,No Financial Incentive
Started | 83 | 84 | 80 | 85 | 82 | 82 | 84 | 82 | 80 | 81 | 81 | 80 | 82 | 85 | 82 | 83
Completed | 79 | 78 | 73 | 82 | 82 | 81 | 81 | 80 | 74 | 79 | 79 | 78 | 78 | 84 | 80 | 78
Not Completed | 4 | 6 | 7 | 3 | 0 | 1 | 3 | 2 | 6 | 2 | 2 | 2 | 4 | 1 | 2 | 5
Not completed — Death | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 6 | 5 | 3 | 0 | 0 | 3 | 1 | 5 | 1 | 2 | 1 | 3 | 0 | 2 | 4
Not completed — Incarcerated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-Call, Patch, SmokefreeTXT, Financial Incentive | 1-Call, Patch, SmokefreeTXT, No Financial Incentive | 1-Call, Patch, No SmokefreeTXT, Financial Incentive | 1-Call, Patch, No SmokefreeTXT, No Financial Incentive | 1-Call, Patch+Loz, SmokefreeTXT, Financial Incentive | 1-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive | 1-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive | 1-Call, Patch+Loz, No SmokefreeTXT, No Financial Incentive | 4-Call, Patch, SmokefreeTXT, Financial Incentive | 4-Call, Patch, SmokefreeTXT, No Financial Incentive | 4-Call, Patch, No SmokefreeTXT, Financial Incentive | 4-Call, Patch, No SmokefreeTXT, No Financial Incentive | 4-Call, Patch+Loz, SmokefreeTXT, Financial Incentive | 4-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive | 4-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive | 4-Call, Patch+Loz, No SmokefreeTXT,No Financial Incentive | Total
Number analyzed (Participants) | 83 | 84 | 80 | 85 | 82 | 82 | 84 | 82 | 80 | 81 | 81 | 80 | 82 | 85 | 82 | 83 | 1316
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.24 (12.36) | 52.82 (11.00) | 55.04 (10.34) | 52.55 (11.36) | 53.43 (12.45) | 51.15 (11.79) | 53.73 (11.08) | 54.12 (11.84) | 52.11 (13.03) | 51.78 (12.58) | 53.49 (12.06) | 54.25 (12.26) | 52.80 (12.25) | 54.41 (12.27) | 53.40 (11.75) | 53.81 (12.23) | 53.13 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender was missing for 2 randomized participants
  Participants
    number analyzed (Participants) | 83 | 84 | 80 | 85 | 82 | 81 | 84 | 82 | 80 | 81 | 81 | 80 | 82 | 85 | 81 | 83 | 1314
    Female | 46 | 51 | 47 | 47 | 48 | 48 | 48 | 48 | 49 | 45 | 46 | 45 | 49 | 49 | 48 | 47 | 761
    Male | 37 | 33 | 33 | 38 | 34 | 33 | 36 | 34 | 31 | 36 | 35 | 35 | 33 | 36 | 33 | 36 | 553
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 5 | 1 | 1 | 2 | 4 | 4 | 2 | 4 | 5 | 0 | 3 | 6 | 3 | 3 | 49
  Not Hispanic or Latino | 80 | 81 | 75 | 84 | 81 | 79 | 80 | 77 | 78 | 73 | 75 | 80 | 79 | 79 | 78 | 80 | 1259
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2 | 3 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 14
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Black or African American | 22 | 20 | 19 | 23 | 22 | 18 | 25 | 21 | 22 | 22 | 22 | 25 | 22 | 22 | 24 | 20 | 349
  White | 54 | 56 | 52 | 56 | 54 | 55 | 52 | 54 | 54 | 54 | 54 | 52 | 55 | 54 | 53 | 57 | 866
  More than one race | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 6
  Unknown or Not Reported | 6 | 4 | 6 | 3 | 5 | 7 | 6 | 6 | 3 | 4 | 5 | 2 | 5 | 6 | 3 | 5 | 76
Region of Enrollment [Number; unit: participants]
  United States | 83 | 84 | 80 | 85 | 82 | 82 | 84 | 82 | 80 | 81 | 81 | 80 | 82 | 85 | 82 | 83 | 1316

OUTCOME MEASURES:

1. Primary Outcome: 7-Day Point-Prevalence Abstinence
Description: Participants will be coded as abstinent if they self-report no smoking for the past 7 days at the assessment endpoint (6 month follow-up) and provide a saliva sample for cotinine testing with a value of <4 ng/ml. Participants will be considered not abstinent if they are lost to follow-up, report any smoking in the past 7 days, return a saliva sample with cotinine greater than or equal to 4 ng/ml, or fail to return a usable saliva sample.
Time Frame: 6-months
Population: All randomized participants were included in intent-to-treat analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Call, Patch, SmokefreeTXT, Financial Incentive | 1-Call, Patch, SmokefreeTXT, No Financial Incentive | 1-Call, Patch, No SmokefreeTXT, Financial Incentive | 1-Call, Patch, No SmokefreeTXT, No Financial Incentive | 1-Call, Patch+Loz, SmokefreeTXT, Financial Incentive | 1-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive | 1-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive | 1-Call, Patch+Loz, No SmokefreeTXT, No Financial Incentive | 4-Call, Patch, SmokefreeTXT, Financial Incentive | 4-Call, Patch, SmokefreeTXT, No Financial Incentive | 4-Call, Patch, No SmokefreeTXT, Financial Incentive | 4-Call, Patch, No SmokefreeTXT, No Financial Incentive | 4-Call, Patch+Loz, SmokefreeTXT, Financial Incentive | 4-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive | 4-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive | 4-Call, Patch+Loz, No SmokefreeTXT,No Financial Incentive
Number analyzed (Participants) | 83 | 84 | 80 | 85 | 82 | 82 | 84 | 82 | 80 | 81 | 81 | 80 | 82 | 85 | 82 | 83
Participants | 11 | 7 | 8 | 10 | 6 | 10 | 10 | 15 | 4 | 16 | 10 | 7 | 12 | 8 | 16 | 12

ADVERSE EVENTS:
Time Frame: 6 months from target quit date (could be 7 months from study enrollment)
Description: The study team assessed hospitalizations at 26-week follow-up as serious adverse assessments. Non-serious adverse events care were assessed by quitline coaches during quitline care and addressed according to standing quitline protocols.
Arm/Group | 1-Call, Patch, SmokefreeTXT, Financial Incentive | 1-Call, Patch, SmokefreeTXT, No Financial Incentive | 1-Call, Patch, No SmokefreeTXT, Financial Incentive | 1-Call, Patch, No SmokefreeTXT, No Financial Incentive | 1-Call, Patch+Loz, SmokefreeTXT, Financial Incentive | 1-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive | 1-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive | 1-Call, Patch+Loz, No SmokefreeTXT, No Financial Incentive | 4-Call, Patch, SmokefreeTXT, Financial Incentive | 4-Call, Patch, SmokefreeTXT, No Financial Incentive | 4-Call, Patch, No SmokefreeTXT, Financial Incentive | 4-Call, Patch, No SmokefreeTXT, No Financial Incentive | 4-Call, Patch+Loz, SmokefreeTXT, Financial Incentive | 4-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive | 4-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive | 4-Call, Patch+Loz, No SmokefreeTXT,No Financial Incentive
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/84 | 2/80 | 0/85 | 0/82 | 1/82 | 0/84 | 1/82 | 1/80 | 1/81 | 0/81 | 0/80 | 1/82 | 1/85 | 0/82 | 1/83
Serious Adverse Events (participants affected / at risk) | 7/83 | 5/84 | 11/80 | 12/85 | 11/82 | 4/82 | 10/84 | 5/82 | 6/80 | 12/81 | 12/81 | 10/80 | 5/82 | 10/85 | 7/82 | 12/83
Other Adverse Events (participants affected / at risk) | 0/83 | 0/84 | 0/80 | 0/85 | 0/82 | 0/82 | 0/84 | 0/82 | 0/80 | 0/81 | 0/81 | 0/80 | 0/82 | 0/85 | 0/82 | 0/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-Call, Patch, SmokefreeTXT, Financial Incentive (N=83) | 1-Call, Patch, SmokefreeTXT, No Financial Incentive (N=84) | 1-Call, Patch, No SmokefreeTXT, Financial Incentive (N=80) | 1-Call, Patch, No SmokefreeTXT, No Financial Incentive (N=85) | 1-Call, Patch+Loz, SmokefreeTXT, Financial Incentive (N=82) | 1-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive (N=82) | 1-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive (N=84) | 1-Call, Patch+Loz, No SmokefreeTXT, No Financial Incentive (N=82) | 4-Call, Patch, SmokefreeTXT, Financial Incentive (N=80) | 4-Call, Patch, SmokefreeTXT, No Financial Incentive (N=81) | 4-Call, Patch, No SmokefreeTXT, Financial Incentive (N=81) | 4-Call, Patch, No SmokefreeTXT, No Financial Incentive (N=80) | 4-Call, Patch+Loz, SmokefreeTXT, Financial Incentive (N=82) | 4-Call, Patch+Loz, SmokefreeTXT, No Financial Incentive (N=85) | 4-Call, Patch+Loz, No SmokefreeTXT, Financial Incentive (N=82) | 4-Call, Patch+Loz, No SmokefreeTXT,No Financial Incentive (N=83)
Infection prompting hospitalization (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Cardiovascular diagnoses and events (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anemia or bleeding disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diabetes complications, thyroid disorder (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Double vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disease, pancreatitis, ulcer, or injury (e.g., hernia) (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Injury or poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer, biopsy, polyp, or cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Stroke, seizure, aneurysm, or suspected multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pregnancy, delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reaction to new psychiatric medication (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation, bipolar, schizophrenia, anxiety, or alcohol use disorder symptoms (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Kidney disease, or kidney or bladder infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease or need for supplemental oxygen (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Planned orthopedic, gastric, or hernia surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Unknown or other reason for hospitalization (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT03538938/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT03538938/ICF_000.pdf